CLINICAL TRIAL: NCT03846999
Title: Comorbidities and Health Care Services Utilisation Among Long-term Breast Cancer Survivors
Acronym: SURBCAN
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); European Regional Development Fund (Other); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other)
Responsible Party: Principal Investigator, Maria Sala, Head of Evaluation and Quality, MD, PhD, Parc de Salut Mar
Other Study IDs: SURBCAN Project
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; comorbidities; healthcare services research; survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long-term breast cancer survivors: Analyze comorbidities and patterns of use of health services. Describe the specific use of health services in primary care vs. specialized care.
  Analyze comorbidities and patterns of use of health services by tumor characteristics.
- Women without history of cancer: Analyze comorbidities and patterns of use of health services. Describe the specific use of health services in primary care vs. specialized care.

SUMMARY:
The increased likelihood of survival can be explained by numerous factors, such as improvements in breast cancer screening and advances in diagnosis and treatment and aging. This phenomenon is associated with comorbidity due to cancer treatment and external factors like aging or lifestyle. Little is known about how these women follow-up their disease, their pattern of use of health resources and their met and unmet needs. Studying the health needs of these women is a cancer-related priority for Cancer Organizations.The project is aimed at: 1) Describing the comorbidities and patterns of use of primary and specialized care in women who have survived a breast cancer for at least five years; 2) Comparing the comorbidities and patterns of use of long time breast cancer survivors with women without a cancer diagnosis; and 3) Estimating the use of resources in long time survivors of breast cancer adjusted for survival-time and comorbidities.

DETAILED DESCRIPTION:
The general objective of this study is to analyze the pattern of comorbidities and utilization of primary care officers and specialized attention of long-term breast cancer survivors and to compare it with women without history of cancer. Long-term breast cancer survivors are those women who survived for at least five years since de primary breast cancer diagnosis.The use of health care services for long-term breast cancer survivors presents new challenges for health systems in terms of defining the role of each health professional and each level of care in contact with these women during their follow-up.

The SURBCAN Project is an observational study that includes a retrospective cohort of women from five Spanish areas. The study is based on Real World Data from clinical history and tumor registration. Women with a diagnosis of breast cancer and a survival period of ≥ 5 years were identified, as well as those women without a cancer diagnosis and matched by age and area with breast cancer survivors (1:2). N= 21639 women (7241 cases /13,398 controls). Sociodemographic and clinical variables were included. The use of primary care and hospital attention and the presence of comorbidities were assessed during the follow-up period (2012-2016). The basal cohort, the comorbidities and the use of health services were described. Factors associated with use were analyzed through multi-level logistic regression models.

Expected results: Nowadays there are no results of cohort analysis that focus specifically in long-term breast cancer survivors. The SURBCAN study will provide evidence regarding comorbidity patterns and follow-up characteristics. The results will guide the elaboration of new recommendations and the decision making by stakeholders concerned to breast cancer survivor's follow-up.

This project combines the experience from experts groups in health services assessment, and analysis of comorbidities and chronic diseases, belonging to the REDISSEC network.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Women diagnosed with an incident breast cancer during the period from 01/01/2000 until 31/12/2006 who survived for at least 5 years.
* Women who visited at least once the primary health services during follow-up period (01/01/2012 to 31/12/2016).

Exclusion Criteria:

- Unknown diagnostic year

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Long-term breast cancer survivors (women who survived at least 5 years from the diagnosis)
Study Population: Women with a diagnosis of breast cancer (during 2000 until 2006) with a survival period of ≥ 5 years that had a visit with the healthcare services during the period from 2012 to 2016 were identified, as well as those women without a cancer diagnosis and matched by age and area with breast cancer survivors.
Sampling Method: Non-Probability Sample
Enrollment: 21639 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of comorbidities | 5 years of survival
  Number of comorbidities of each woman at five-year survival from breast cancer. Assessed through ICD10.
Frequency of visits to healthcare services | 5 years of survival
  Number of visits to primary care attention or specialised attention done by each women at five-year survival from breast cancer.
Main health provider visited | 5 years of survival
  Leading provider of health services (GP, oncologist, community nurse, oncology nurse, physiotherapist...) of each women at five-year survival from breast cancer.

SECONDARY OUTCOMES:
Frequency of visits to primary care attention | at 5 years of survival
  Number of visits to primary care attention done by each women at five-year survival from breast cancer.
Frequency of visits to specialized care attention | at 5 years of survival
  Number of visits to specialised attention done by each women at five-year survival from breast cancer.
Annual mammogram frequency | 1 year
  Assessment of the percentage of women who have a mammogram every year.

REFERENCES:
- [Derived] Jansana A, Del Cura I, Prados-Torres A, Sanz Cuesta T, Poblador-Plou B, Gimeno Miguel A, Lanzuela M, Ibanez B, Tamayo I, Moreno-Iribas C, Padilla-Ruiz M, Redondo M, Comas M, Domingo L, Diaz-Holgado A, Salamanca FJ, Castells X, Sala M; SURBCAN group. Use of real-world data to study health services utilisation and comorbidities in long-term breast cancer survivors (the SURBCAN study): study protocol for a longitudinal population-based cohort study. BMJ Open. 2020 Sep 9;10(9):e040253. doi: 10.1136/bmjopen-2020-040253. PMID 32912957